CLINICAL TRIAL: NCT06001684
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of IBR854 Cell Injection in Patients With Unresectable Locally Advanced Or Metastatic Solid Tumors
Brief Title: Phase 1 Study of IBR854 in Locally Advanced Or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ning Li, MD, PhD, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBR854-101
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBR854 Cell Injection (Experimental): The minimum initial dose is 3.0×10^9 cells and then escalate to 5.0×10^9 cells and 7.0×10^9 cells. Every 21 days is one cycle, and intravenous infusion is performed on day 1 and day 8 of each cycle.
  Interventions: Biological: IBR854 Cell Injection

INTERVENTIONS:
Biological: IBR854 Cell Injection — The minimum initial dose is 3.0×10^9 cells and then escalate to 5.0×10^9 cells and 7.0×10^9 cells. Every 21 days is one cycle, and intravenous infusion is performed on day 1 and day 8 of each cycle.

SUMMARY:
This study is an open-label, phase I study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of IBR854 cell injection in patients with unresectable, locally advanced, or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is a dose escalation study which adopts the 3+3 dose escalation design protocol. The dose is respectively 3.0×10^9 cells, 5.0×10^9 cells and 7.0×10^9 cells. The administration is performed on day 1 and day 8 of each cycle (21 days). 3-6 subjects will be enrolled at every dose level. The first and second subjects in the same group shall be enrolled at an interval of at least 7 days, for the purpose of ensuring their safety. Only when the dose-limiting toxicity (DLT) of all subjects in the previous dose group was observed can the enrollment of the next dose group get started.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteer to participate in this clinical study, are fully aware of the study and have signed the Informed Consent Form (ICF). Subjects are willing to follow and able to complete all trial procedures.
2. Age: adult at the age of 18-75 (both inclusive), female or male.
3. Subjects with histologically or cytologically confirmed, unresectable, locally advanced or metastatic solid tumors (which can be diagnosed with the use of tumor markers in combination with imaging for specific advanced tumors, such as liver cancer) who have no current standard of care.
4. Eastern Cooperative Oncology Group (ECOG) score ≤2 and expected survival time >3 months.
5. According to the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 criteria, the subjects have at least one target lesion (non-lymph node lesion with major diameter ≥ 1.0cm or lymph node lesion with minor diameter ≥ 1.5 cm). A lesion that is within the field of previous radiotherapy could not be considered a target unless there is radiographic evidence of progression.
6. Organ function during screening should meet the following criteria:

   * Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet (PLT) ≥75×10^9/L; Hemoglobin (Hb)≥80g/L (no blood transfusion or hematopoietic stimulator treatment within 7 days).
   * Alanine aminotransferase (ALT)≤3×ULN (Patients with liver metastasis: ≤5×ULN); Aspartate aminotransferase (AST)≤3×ULN (Patients with liver metastasis: ≤5×ULN);
   * Creatinine (Cr) ≤2× ULN; Creatinine clearance (Ccr) (to be calculated only when Cr > 2× ULN) > 50ml/min (Cockcroft-Gault formula);
   * Activated partial thrombin time (APTT) ≤1.5×ULN, International normalized ratio (INR) ≤1.5×ULN (Patients with anticoagulants: ≤ 2.5×ULN).
7. Subjects of reproductive age and their partners should agree to have no family planning and to use effective contraceptive methods for 6 months from signing the ICF until the last dose of the study drug is administered.

Exclusion Criteria:

1. Have received systemic antitumor therapy within 4 weeks or five half-lives of the drug (whichever is longer) before the first dose of the study drug: Systemic chemotherapy (2 weeks for oral fluorouracil, 6 weeks for mitomycin C and nitrosoureas), endocrine therapy, targeted therapy (2 weeks or 5 half-life for small molecule targeted therapy, whichever is longer), immunotherapy, radical radiotherapy, tumor embolization, Chinese herbal medicine for anti-tumor indications, etc. Or received palliative radiotherapy within 2 weeks before the first dose.
2. Toxic effects from previous antitumor therapy have not returned to grade 1 or less (other than alopecia or fatigue).
3. Any prior adoptive cellular immunotherapy.
4. Active brain metastases (one of the following criteria: clinical symptoms; A new diagnosis; Progression after previous local treatment).
5. Have undergone major organ surgery within 4 weeks prior to their first use of the study drug, or required elective surgery during the study period.
6. Long-term (≥ 3 days) treatment with a glucocorticoid (prednisone > 10 mg per day or equivalent) or another immunosuppressive agent is anticipated to be required during the study. Inhaled or topical steroid hormones are allowed in subjects without active autoimmune disease
7. Have received a live or attenuated vaccine within 4 weeks before the first dose or plan to receive a live or attenuated vaccine during the study period.
8. Have severe infections that cannot be controlled.
9. Active hepatitis B, hepatitis C virus infection or HIV infection.
10. Have undergone an allogeneic bone marrow transplant or other organ transplant.
11. Have active autoimmune diseases or have had autoimmune diseases that are likely to recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, psoriasis, etc.). Except in the following cases: type 1 diabetes that was well controlled with hormone replacement therapy, hypothyroidism, skin conditions that did not require systemic therapy (e.g., vitiligo), and other conditions that were well controlled and that the investigator determined were less likely to recur (e.g., childhood asthma in remission).
12. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    * There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia, and Ⅱ-Ⅲ degree atrioventricular block, which need clinical intervention;
    * Prolonged QT interval corrected with Fridericia's method (QTcF) (>450 ms in men; >470 ms for women)
    * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurring within 6 months before the first administration;
    * Patients with heart failure or left ventricular ejection fraction (LVEF) < 50% in the New York Heart Association (NYHA) classification ≥II;
    * Hypertension beyond clinical control.
13. Clinically significant chronic obstructive pulmonary disease or other moderate to severe chronic respiratory disease developed within 6 months.
14. Have other malignant tumors in the past 3 years, excluding skin basal cell carcinoma, ductal carcinoma in situ and cervical carcinoma in situ with a radical surgery.
15. Pregnant or lactating women.
16. Have mental disorders or a history of alcohol, drug or drug abuse within one year.
17. Have participated in other clinical trials and received any unmarketed investigational drug or treatment within 4 weeks prior to first use of the study drug.
18. Allergic to the main components of the study drug.
19. The investigator considered that the subjects had a history of other serious systemic diseases or other reasons that made them unsuitable for the study.
20. Unsuitable for participation in this study considered by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | From day1 to day 21
  To collect dose limiting toxicities (DLTs) occurring within 21 days after the first dose
The incidence and severity of adverse events (AEs) | From day 1 to day 90 after the first dose
  To evaluate the safety of IBR854 cell injection

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  To determine the anti-tumor effectivity of IBR854 cell injection
Disease control rate (DCR) | 1 year
  To determine the anti-tumor effectivity of IBR854 cell injection
Duration of remission (DOR) | 1 year
  To determine the anti-tumor effectivity of IBR854 cell injection
Progression-free survival (PFS) | 1 year
  To determine the anti-tumor effectivity of IBR854 cell injection
Overall survival (OS) | 1 year
  To determine the anti-tumor effectivity of IBR854 cell injection
The number of IBR854 cells | 1 year
  Blood samples will be collected at specified time points to detect the number of IBR854 cells in peripheral blood
Anti-CAR antibodies | 1 year
  Blood samples will be collected at specified time points to detect anti-CAR(anti-5T4 mAb) antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No